CLINICAL TRIAL: NCT07047365
Title: A Randomized, Open-label, Parallel-controlled, Multicenter Phase III Clinical Study Evaluating TQB2930 Combined With Investigator's Choice of Chemotherapy Versus Trastuzumab Combined With Investigator's Choice of Chemotherapy in the Treatment of HER2-Positive Advanced Breast Cancer
Brief Title: TQB2930 Injection for the Treatment of HER2-positive Advanced Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2930-III-01
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2930+ chemotherapy (Experimental): Subjects will receive TQB2930 injection in combination with chemotherapy agents on Day 1 (D1) of each cycle. TQB2930 will be administered at a dose of 30 mg/kg every 3 weeks (Q3W), Each treatment cycle lasts 21 days.
  Interventions: Drug: TQB2930+ chemotherapy
- Trastuzumab+ chemotherapy (Active Comparator): Subjects will receive trastuzumab in combination with chemotherapy agents on Day 1 (D1) of each cycle. The initial dose of trastuzumab is 8 mg/kg, followed by a maintenance dose of 6 mg/kg administered every 3 weeks (Q3W), Each treatment cycle lasts 21 days.
  Interventions: Drug: Trastuzumab+ chemotherapy

INTERVENTIONS:
Drug: TQB2930+ chemotherapy — TQB2930 injection is a HER2 bispecific antibody drug； Chemotherapy: Capecitabine Tablets, Gemcitabine Hydrochloride for Injection, Vinorelbine Tartrate Injection and Eribulin Mesylate Injection are Chemotherapy Drugs.
  Arms: TQB2930+ chemotherapy
Drug: Trastuzumab+ chemotherapy — Trastuzumab is a HER2-specific targeted drug； Capecitabine Tablets, Gemcitabine Hydrochloride for Injection, Vinorelbine Tartrate Injection and Eribulin Mesylate Injection are Chemotherapy Drugs.
  Arms: Trastuzumab+ chemotherapy

SUMMARY:
TQB2930 is a HER2 bispecific antibody drug. This study aims to evaluate the efficacy and safety of TQB2930 combined with investigator's choice of chemotherapy versus trastuzumab combined with investigator's choice of chemotherapy in subjects with HER2-positive advanced breast cancer who have received at least two prior lines of anti-HER2 therapy in the advanced station.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign the informed consent form;
* Age: 18-75 years (at time of signing Informed Consent Form (ICF); Eastern Cooperative Oncology Group (ECOG) performance status ≤1; estimated life expectancy >3 months;
* Cytologically or histologically confirmed Human Epidermal Growth Factor Receptor 2 (HER2)-positive recurrent or metastatic breast cancer;
* Received ≥2 prior lines of anti-HER2 targeted therapy in the advanced setting;
* At least one measurable lesion meeting Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) criteria (excluding brain lesions);
* Willing to receive one of the investigator-selected chemotherapy regimens;
* Adequate organ function;
* Female subjects of childbearing potential must agree to use effective contraception (e.g., Intrauterine Device (IUD), oral contraceptives, or condoms) during the study and for 6 months after study completion.

Exclusion Criteria:

* Concurrent Diseases and Medical History:

  * Other malignancies within 5 years before randomization or concurrent malignancies (except adequately treated non-melanoma skin cancer, in situ cervical cancer, or other cancers with curative treatment and no recurrence for ≥3 years);
  * Uncontrolled toxicities (>CTCAE Grade 1) from prior therapies (excluding alopecia);
  * Major surgery, open biopsy, or significant traumatic injury within 28 days before randomization;
  * Non-healing wounds or fractures;
  * Arterial/venous thromboembolic events within 6 months before randomization;
  * History of drug abuse or psychiatric disorders that may affect compliance;
  * Poorly controlled hypertension (e.g., Systolic Blood Pressure (SBP) >160 mmHg despite treatment);
  * ≥Grade 2 myocardial ischemia/infarction, arrhythmias, or congestive heart failure (New York Heart Association （NYHA）Class ≥II);
  * Active or uncontrolled severe infections (≥CTCAE Grade 2);
  * Known chronic hepatitis B;
  * Active syphilis infection;
  * Renal failure requiring hemodialysis/peritoneal dialysis;
  * Immunodeficiency disorders (e.g., Human Immunodeficiency Virus (HIV) ;
  * Poorly controlled diabetes;
  * Urine protein ≥++ on dipstick with 24-hour urine protein >1.0 g;
  * Epilepsy requiring medication.
* Tumor-Related Conditions and Treatments:

  * Chemotherapy, radiotherapy, or immunotherapy within 4 weeks before randomization (or within 5 half-lives of prior drugs, whichever is shorter);
  * Chinese herbal medicines with approved antitumor indications (per National Medical Products Administration (NMPA) labeling) within 2 weeks;
  * Severe Bone Lesions from bone metastases;
  * Untreated brain metastases, Leptomeningeal metastases, or carcinomatous meningitis;
  * Prior HER2-targeted therapy-induced Left Ventricular Ejection Fraction (LVEF) decline to <50% or absolute reduction >15%;
  * Uncontrolled or symptomatic Hypertension requiring ongoing bisphosphonates;
  * Uncontrolled cancer-related pain;
  * Existed Lymphangitis Carcinomatosa or uncontrolled effusions;
  * Use of Immunosuppressant or systemic corticosteroids (≥10 mg/day prednisone equivalent) within 2 weeks.
* Severe hypersensitivity to monoclonal antibodies;
* Participation in other antitumor clinical trials with investigational drugs within 4 weeks before randomization;
* Any condition deemed by the investigator to jeopardize subject safety or study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to IRC-assessed Disease Progression(PD), approximately 1 years
  Independent Imaging Review Committee (IRC)-assessed PFS

SECONDARY OUTCOMES:
PFS assessed by Investigator | Baseline up to Investigator-Assessed investigator, approximately 1 years
  PFS assessed by Investigator
Overall survival (OS) | From date of the first dose until the date of death from any cause, up to approximately 2 years
  From randomization to the time of death from any cause.
Duration of Response (DOR) | From date of the first dose until the date of first documented progression or date of death from any cause, up to approximately 2 years
  Subjects with best overall response of complete response (CR) or partial response (PR) per RECIST 1.1 criteria.
Proportion of subjects achieving partial response (PR) | From the date of first documented tumor response to the date of first documented disease progression or death from any cause (whichever occurs first), up to approximately 1 years
  Subjects with partial response (PR) per RECIST 1.1 criteria.
Objective Response Rate (ORR) | From the date of first documented tumor response to the date of first documented disease progression or death from any cause (whichever occurs first), up to approximately 1 years
  Percentage of subjects achieving complete response (CR) or partial response (PR) per RECIST 1.1 criteria.
Clinical Benefit Rate (CBR) | From the date of first documented tumor response to the date of first documented disease progression or death from any cause (whichever occurs first) , up to approximately 1 years
  Proportion of subjects with best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD) lasting ≥24 weeks per RECIST 1.1 criteria.
Adverse event rate | From baseline until 90 days after the last dose or initiation of new antitumor therapy, whichever occurs first
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Plasma concentration of TQB2930 | Within 60 minutes before dosing on Cycle 1 Day 1, Cycle 4 Day 1, Cycle 7 Day 1, and Cycle 12 Day 1; and within 30 minutes after dosing on Cycle 4 Day 1 and Cycle 7 Day 1, each cycle is 21 days
  Serum concentrations of TQB2930 in subjects after administration in the treatment group.
Anti-Drug Antibody (ADA) Positivity Rate | Within 60 minutes before dosing on Cycle 1 Day 1, Cycle 4 Day 1, Cycle 7 Day 1, and Cycle 12 Day 1; and within 90 days after the last dose, each cycle is 21 days
  Anti-drug antibody (ADA) positivity in post-dose blood samples from subjects in the treatment group.
Anti-Drug Antibody (ADA) Positivity Rate | Within 60 minutes before dosing on Cycle 1 Day 1, Cycle 4 Day 1, Cycle 7 Day 1 , and Cycle 12 Day 1; and within 90 days after the last dose, each cycle is 21 days
  Neutralizing antibody (NAb) testing performed when anti-drug antibodies (ADAs) were detected in post-dose blood samples from the treatment group.

CONTACTS AND LOCATIONS:
Locations (69):
- China (69):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital( The First Affiliated Hospital of USTC), Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Chong Qing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fuzhou First Generel Hospital Affiliated with Fujian Medical University, Fuzhou, Fujian
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Sun Yat - sen University Cancer Center, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Affiliated Cancer Hospital of Guangxi Medical Universit, Nanning, Guangxi
  - The Affiiated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiamusi Tuberculosis Hospital (Jiamusi Tumor Hospital), Jiamusi, Heilongjiang
  - Mudanjiang Cancer Hospital, Mudanjiang, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jingmen People's Hospital, Jingmen, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Zhangjiajie People's Hospital, Zhangjiajie, Hunan
  - JiangSu Cancer Hosipital, Nanjing, Jiangsu
  - The Affiliated Sir Run Run Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhangjiagang First People's Hospital, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital Of Dalian University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Bao Ji Central Hospital, Baoji, Shaanxi
  - 3201 Hospital, Hanzhong, Shaanxi
  - The Second Affiliated Hospital Of Xi'an Jiaotong University (Xibei Hospital), Xi'an, Shaanxi
  - Xijing Hospital of Air Force Military Medical University, Xi'an, Shaanxi
  - Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute,Shandong Cancer Hospital), Jinan, Shandong
  - Linyi cancer Hospital, Linyi, Shandong
  - Weifang People'S Hospital, Weifang, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - The Second People's Hospital of Yibin City, Yibin, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Affiliated Tumor Hospital, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Ningbono.2Hospitai, Ningbo, Zhejiang
  - The First Affiliated Hospial of Ningbo University, Ningbo, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang